CLINICAL TRIAL: NCT05412810
Title: Oxidative Lipidomic Biomarkers During Mechanical Ventilation in Critically Ill Patients (OXY-BAL).
Acronym: OXY-BAL
Status: Recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Sonal Pannu, Principal Investigator, Ohio State University
Other Study IDs: 2018H0302
Record Dates: First submitted 2022-04-15; First posted 2022-06-09 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Mechanical Ventilation Complication; Hyperoxia
MeSH Terms: conditions — Hyperoxia | interventions — Oxygen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — All consenting patients will have an additional 5 ml bronchoalveolar fluid collected during the procedure. Additionally, 5 cc blood will also be collected to correlate with the BAL samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Oxygen exposures: mechanically ventilated patients with atleast 1.5 hours of FiO2 exposure of 50% or more
  Interventions: Other: oxygen

INTERVENTIONS:
Other: oxygen — oxygen exposure of more than 50% for 1.5 hours

SUMMARY:
The aim of this study is to identify and determine the levels of oxidized lipids and lipid mediators following exposure to oxygen supplementation during mechanical ventilation by oxidative lipidomics. The investigators will include patients with mechanical ventilation and have received FiO2=>0.5 atleast 90 minutes and collected two sequential mini bronchoalveolar lavage on them 24 hours apart. Mass Spectrometry Lipid chromatography will be conducted and clinical data will be analyzed.

DETAILED DESCRIPTION:
This proposal will elucidate an approach for precise and safe oxygenation levels and correlation with the oxidative lipid biomarker profile of optimal oxygenation. The aim of this study is to identify and determine the levels of oxidized lipids and lipid mediators following exposure to oxygen supplementation during mechanical ventilation by oxidative lipidomics. Alveolar cellular membrane and lung lining fluid are the primary targets of therapeutic oxygen and comprised of proteins, cholesterol, and lipids. Among these components, lipids are more susceptible to oxidation producing downstream mediators that facilitate inflammatory and pro-fibrotic pathways. Polyunsaturated Fatty Acids (PUFAs) account for 30% of the lipid components and contain n-3 fatty acids (i.e eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA)) and n-6 fatty acids ( arachidonic acid (AA) and Dihomo-γ-linolenic acid (DGLA)). In the presence of reactive oxygen species and activation of the metabolic enzymes (e.g. cyclooxygenases and lipoxyegenases), n-3 and n-6 PUFAs undergo peroxidation to form "oxidized forms" and are further metabolized into numerous proinflammatory and proresolving lipid mediators. Many of these lipid mediators (Prostaglandin E2, PGE2; 11-hydroxy--eicosatetraenoic acid 11-HETE, 5-hydroxy-eicosapentaenoic acid 5-HEPE) perpetuate inflammatory mechanisms known to mediate HALI45. Additionally, some of these mediators known as specialized proresolving mediators (SPMs) dampen inflammation while promoting pro-resolution actions on tissue inflammation after injury (e.g maresins, Resolvin D5). Lipidomics is one of the most sensitive approaches for studying lipid profiles in clinical research. Given the access to lung samples (bronchoalveoar fluid; BALF) in the setting of acute hypoxemic respiratory failure in the ICU, this provides strong rationale to utilize this largely unexplored method to guide clinical practice of optimal oxygenation goals.

We propose a prospective cohort study to evaluate oxidized lipid biomarkers in the BALF of patients with acute hypoxemic respiratory failure. Inclusion criteria are 1) Adults ≥ 18 years with acute hypoxemic respiratory failure 2) with expected MV => 48 hours. Exclusion criteria are 1) MV for procedures like EGD, bronchoscopy , colonoscopy;2) Chronic respiratory failure prior to admission; 3) Hemoptysis, diffuse alveolar hemorrhage; 3) Primary team prohibits bronchoscopy for a specific clinical indication or safety; 4) Medication use such as N acetyl cysteine; aspirin, fish oil supplements. Control subjects will be those with MV without acute hypoxemic or hypercarbic respiratory failure (e.g. MV due to stroke or seizures). Informed consent will be taken. All consenting patients will have a two sequential BALF collections by collected from patients on day 1 (≤6 hours of MV if initial FiO2 use is ≥0.5 for 90 minutes) and day 2 (≥48 hours after the first BALF). We have specifically chosen these time points because Day 1 will allow us to define initial oxidized n-6 PUFA precursor levels and their relationship to clinical outcomes. Since markers of lipid peroxidation are at the highest on Day 2, these Day 2 samples will allow us to define the trajectory of oxidized n-6 PUFA and associate these with clinical outcomes.

Following the BAL collection, it will be stored at -80 and Liquid chromatography-mass spectrometry will be used for oxidative lipidomic analysis of ~130 oxidized lipid species. Patient data will be abstracted from the chart at time of enrollment. Clinical data variables will include: 1) demographics; 2) medical history 3) hourly FiO2 and SpO2 4) Sequential Organ Failure Assessment (SOFA) scores for disease severity; 5) daily arterial blood gas for PaO2/FiO2 ratio 6) daily vital signs 7) clinical laboratory studies (blood counts for hemoglobin, electrolyte panel, lactic acid levels; 8) medications; and 9) outcomes measures (ventilator-free days, survival). More importantly, we will note co-morbidities and treatment related variables that may independently modify oxidized lipids and serve as confounders. Such smoking status, active lung or breast cancer, quantity and nature of tube feeds, use of propofol (a lipid emulsion) for sedation, and utilization of immune modulators such as steroids, will be noted and will be adjusted for univariate and multivariate analysis.

ELIGIBILITY:
Inclusion Criteria:

• Adults age => 18 and needing Mechanical ventilation in Intensive Care unit expected atleast for 48 hours

Exclusion Criteria:

* 1.Mechanical ventilation, only needed for performing procedures- bronchoscopy, esophagogastroduodenoscopy, colonoscopy, or others
* 2)Chronic respiratory failure prior to admission;
* 3)Hemoptysis or diffuse alveolar hemorrhage
* 4)Medication use such as N acetyl cysteine; aspirin, fish oil supplements.
* 5)Primary team prohibits bronchoscopy for a specific clinical indication or safety;

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will include all patients who are mechanically ventilated and age above >=18 years. We will consent a patient if a bronchoalveolar lavage via fiber optic bronchoscopy (BAL) or through tracheal catheter (mini - BAL) is indicated for clinical care up to 72 hours since intubation and mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Oxidized n6-PUFAs (Poly Unsaturated Fatty Acids) | days 1, and 2
  Polyunsaturated fatty acids will be measured by mass spectrometry and compared in patients with optimized vs liberal oxygenation with moderated t tests
Oxidized n3-PUFAs (Poly Unsaturated Fatty Acids) | days 1, and 2 of mechanical ventilation
  Polyunsaturated fatty acids will be measured by mass spectrometry and compared in patients with optimized vs liberal oxygenation with moderated t tests

SECONDARY OUTCOMES:
Pro- inflammatory mediators-Prostaglandin E2, PGE2; 11-hydroxy--eicosatetraenoic acid 11-HETE, 5-hydroxy-eicosapentaenoic acid 5-HEPE | days 1, and 2 of mechanical ventilation
  lipid mediators will be measured by mass spectrometry and compared in patients with optimized vs liberal oxygenation with moderated t tests
Correlation of oxidized lipid and lipid mediators to degree of oxygenation and oxygen delivery | From enrollment to liberation from mechanical ventilation or death whichever occurs earlier assessed upto 90 days
  AA, DGLA and lipid mediators levels in each category will be correlated to ventilator-free days using an analysis of covariance (ANCOVA) model. Other significant co variates will be assessed in multivariate logistic regression. Ventilator free days will be calculated

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States